CLINICAL TRIAL: NCT07352774
Title: Effects of Laughter Therapy on Respiratory Functions and Geriatric Pain in Elderly Individuals
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Nisa Nur AKBAL, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraU-Nrs-NA-01; TYL-2025-4407 (Other Grant/Funding Number: Ankara University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2025-12-24; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Elderly; Respiratory Function; Pain
Keywords: Laughter Therapy; Respiratory Function; Pain; Elderly
MeSH Terms: conditions — Respiratory Aspiration; Pain | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Two randomly controlled groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): A pulmonary function test and a geriatric pain scale were administered to this group. No intervention was made. A pulmonary function test and a geriatric pain scale were administered again one month later.
- Laughter Therapy (Experimental): A pulmonary function test and a geriatric pain scale were administered to this group and this group received laughter therapy 8 times in total, twice a week for 1 month. Respiratory function test and geriatric pain scale were applied before the intervention.
  Interventions: Behavioral: Laughter Therapy

INTERVENTIONS:
Behavioral: Laughter Therapy — A laughter therapy session lasts 45-50 minutes. It includes 10 minutes of warm-up exercises, 15 minutes of breathing exercises, and 15 minutes of laughter exercises. It concludes with a 5-10-minute meditation.
  Arms: Laughter Therapy

SUMMARY:
This study aimed to evaluate the effects of laughter therapy on respiratory functions and geriatric pain in elderly individuals.

DETAILED DESCRIPTION:
Structural and functional changes occur with aging and are seen as a decrease in body functions. One of the body systems of aging is the respiratory system capacity. Aging causes the lung tissue to lose elasticity, the respiratory muscles to weaken, and the gas exchange to not be carried out effectively, causing a decrease in respiratory capacity. Therefore, it causes shortness of breath in individuals, an increase in the risk of climate change, and a decrease in the quality of life. Changes in body systems also cause chronic pain in the elderly. Pain-related loss of strength, functional losses, and multiple drug use are observed. Complementary treatment methods can be used against these changes caused by aging, to reduce the problems of old age and for healthy aging. The aim of these therapies is to increase the respiratory capacity of the elderly and the intensity of geriatric pain.

The universe of the study consists of individuals who are members of a Retirement Club affiliated to Ankara Metropolitan Municipality and who do not have any visual, auditory, mental or orthopedic disabilities, aged 60 and over and who agreed to participate in the study. 64 individuals who meet the inclusion criteria constitute the sample of this study. The sample will be randomly selected from the true random number selector (https://www.random.org/) website. Random selections will be planned as a sequential intervention and a control group, respectively. Selection will continue until the sample size is completed. As part of the pre-test, an introductory information form, Respiratory Function Test, oxygen saturation measurement with pulse oximeter, respiration count and Geriatric Pain Scale will be applied to the individuals in the intervention and control groups. The intervention group will receive 8 sessions of laughter therapy twice a week for 4 weeks. No intervention will be applied to the control group. As part of the post-test, the intervention and control groups will be applied; Respiratory Function Test, oxygen saturation measurement with pulse oximetry, respiratory count and Geriatric Pain Scale will be applied. Research data will be analyzed using the Statistical Package for Social Sciences (SPSS) 25.0 program.

Laughter therapy is a complementary medicine technique that combines laughter for no reason and breathing exercises. Laughter therapy is a free, accessible, effective and enjoyable intervention for individuals. Laughter therapy has been accepted as a nursing intervention in the Nursing Intervention Classification at the international level. Laughter therapy increases lung capacity and ensures effective gas exchange thanks to the breathing exercises it contains. It is thought that laughter therapy, which includes breathing exercises, can also provide positive developments in respiratory parameters. Laughter therapy is thought to be an effective intervention in improving respiratory functions and reducing pain.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Dikmen Retirees' Club, who do not accept to leave, are 60 years of age or older, have any work, visual, mental or orthopedic disability that would prevent them from participating in the sections, including those who smoke and use alcohol.

Exclusion Criteria:

* Being under 60 years of age and having conditions that prevent the application of laughter therapy (having had abdominal surgery in the last three months, glaucoma, hernia and epilepsy), smoking and drinking alcohol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Geriatric Pain Scale | 4 weeks
  The original scale, called the Geriatric Pain Measure, is a twenty-four-item multidimensional scale developed by Ferrell and colleagues in 2000. The scale adapted for Turkish has five dimensions, as in the original. It includes subscales for pain withdrawal (items 19, 20, 22, and 23), pain intensity (items 1, 2, 3, 4, 5, and 6), pain with movement (items 9, 10, 11, and 12), pain due to strenuous activities (items 7, 8, 18, 21, and 24), and pain due to other activities (items 13, 14, 15, 16, and 17). The scale includes two open-ended questions (items 19 and 20). These questions are scored from 0 to 10. For the other 22 items, each "Yes" response is summed and multiplied by 2.38. The total possible score ranges from 0 to 100. A score between 0 and 29 indicates mild pain, a score between 30 and 69 indicates moderate pain, and a score of 70 or above indicates severe pain. The total Cronbach's alpha value for the scale is 0.85.
Forced Vital Capasity: FVC | 4 weeks
  Mean Change from Baseline in Forced Vital Capacity (FVC) at Week 4. FVC is the total amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. It will be used to assess the improvement or stabilization of total lung volume.
  Unit of Measure: Liters (L)
Forced Expiratory Volume in 1 Second: FEV1 | 4 weeks
  Mean Change from Baseline in Forced Expiratory Volume in 1 Second at week 4. The absolute volume of air exhaled during the first second of the forced vital capacity maneuver. The highest value from three acceptable maneuvers will be recorded in liters (L).
FEV1/FVC Ratio | 4 weeks
  Mean Change from Baseline in FEV1/FVC Ratio at Week 4. This ratio (Tiffeneau-Pinelli index) represents the percentage of vital capacity a person can deliver in the first second of a forced exhalation. It is used to differentiate obstructive and restrictive lung patterns.
  Unit of Measurement: Percentile
Peak Expiratory Flow: PEF | 4 weeks
  Mean Change from Baseline in Peak Expiratory Flow (PEF) at Week 4. PEF measures the maximum exhalation rate.
  Unit of Measurement: Liters/minute (L/min)
Forced Expiratory Flow: FEF 25-75 | 4 weeks
  Change from Baseline in Forced Expiratory Flow Between 25% and 75% of Vital Capacity (FEF 25-75%) at Week 4. This measure reflects the flow rate during the middle half of the FVC maneuver and is a sensitive indicator of small airway function.
  Unit of Measure: Liters per second (L/sec)

SECONDARY OUTCOMES:
Oxygen Saturation | 4 weeks
  Mean Change from Baseline in Oxygen Saturation at Week 4 Oxygen saturation indicates the oxygenation level of the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özlem Öztürk, ASSOCİATE PROFESSOR, Study Director — ANKARA UNİVERSİTY
Locations (1):
- Ankara University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available beginning 6 months after publication of the study results and for a period of 5 years.
Access Criteria: Researchers must provide a formal request and a statistically sound proposal to access the data. Requests will be reviewed by the principal investigator.

DOCUMENTS (2):
  • Study Protocol (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT07352774/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT07352774/SAP_001.pdf